CLINICAL TRIAL: NCT02285582
Title: International Rare Histiocytic Disorders Registry (IRHDR)
Acronym: IRHDR
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Oussama Abla, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000045224
Record Dates: First submitted 2014-11-03; First posted 2014-11-07 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Rare Histiocytic Disorders (RHDs); Erdheim-Chester Disease (ECD); Rosai-Dorfman Disease (RDD); Xanthogranuloma Family (XG); Indeterminate Dendritic Cell Histiocytosis; Malignant Histiocytic Neoplasm (MHN); ALK-positive Histiocytosis; Mixed Histiocytosis (MXH); Multicentric Reticulohistiocytoma (MRH); Necrobiotic Xanthogranuloma (NX)
MeSH Terms: conditions — Erdheim-Chester Disease; Histiocytosis, Sinus; Necrobiotic Xanthogranuloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Registry study — No intervention.

SUMMARY:
The rare histiocytic disorders (RHDs) are characterized by the infiltration of one or more organs by non-LCH histiocytes. They can range from localized disease that resolves spontaneously, to progressive disseminated forms that can be sometimes life-threatening. Since they are extremely rare, there is limited understanding of their causes and best treatment options. Physicians, patients and parents of children with RHDs frequently consult members of the Histiocyte Society regarding the best management of these disorders. Very often, no specific recommendation can be made due to the lack of prospective outcome data, or even large retrospective case series. The creation of an international rare histiocytic disorders registry (IRHDR) could facilitate a uniform diagnosis of the RHDs, as well as the collection and analysis of the clinical, epidemiological, treatment and survival data of patients with RHD. The registry may also lead to future therapeutic recommendations, provide a framework for future clinical trials and create excellent research opportunities.

DETAILED DESCRIPTION:
Histiocytoses are rare diseases caused by an excess of cells called Histiocytes, which can infiltrate the skin, bones, lungs, liver, spleen and the central nervous system. These disorders can range from localized involvement that resolves spontaneously, to progressive disseminated forms that can be debilitating and sometimes life-threatening. The rare histiocytic disorders (RHD), or non-Langerhans cell disorders, are a diverse group of disorders defined by the accumulation of histiocytes that do not meet the criteria for Langerhans cell histiocytosis (LCH) or hemophagocytic lymphohistiocytosis (HLH). They include: Juvenile xanthogranuloma family, Erdheim-Chester disease, Multifocal Reticulohistiocytosis, Rosai-Dorfman disease and the Malignant Histiocytoses. Since they are so rare, there is limited understanding of their causes and treatments. Physicians, patients and parents of children with rare histiocytoses frequently consult members of the Histiocyte Society on the management of these disorders. Very often, no specific recommendation about treatment can be made due to the lack of prospective outcome data for these rare entities. The creation of an International Rare Histiocytic Disorders Registry (IRHDR) will facilitate a uniform diagnosis of the RHD's, as well as the collection and analysis of the clinical, epidemiological, treatment and survival data of patients with RHD. The registry will also provide expert pathology reviews and may lead to future therapeutic recommendations. Furthermore, the IRHDR can provide a framework for future clinical trials, thus, creating excellent research opportunities. Lastly, a de-identified link between clinical data and companion biology studies can potentially be accomplished in the future through the IRHDR. This may further help in understanding the etiology of these rare diseases, as well as identifying potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. Any age at diagnosis.
2. Diagnosis of a rare histiocytic disorder, established before or after the opening of the registry.
3. Cases diagnosed from January - 01- 1995 until the present time and prospectively.
4. Signed informed consent by a patient, or parent/legal guardian.
5. Cognitively impaired patients can be included after consent by legal guardian/parent.
6. Deceased patients can be included if they are contacted at least 6 months after the death of their child and not on their child's birthday or anniversary of death.

Exclusion Criteria:

1. Informed consent has not been signed.
2. Diagnosis other than RHD.
3. Cases diagnosed before the year 1995.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rare Histiocytic Disorders:
  1. Xanthogranuloma Family (XG)
     * Cutaneous
     * Benign cephalic histiocytosis (BCH)
     * Generalized eruptive histiocytosis (GEH)
     * Progressive nodular histiocytosis (PNH)
     * Xanthoma disseminatum (XD)
     * Giant XG
     * Reticulohistiocytoma
     * Ocular
     * Systemic
  2. Erdheim-Chester Disease (ECD)
  3. Rosai-Dorfman disease (RDD)
     * Single system
     * Nodal
     * Extranodal
     * Skin
     * CNS
     * Bone
     * Orbit
     * Other
     * Multisystemic
  4. Indeterminate Dendritic Cell Histiocytosis
  5. Malignant Histiocytic Neoplasm (MHN)
     * Histiocytic
     * Langerhans cell
     * Interdigitating dendritic cell
     * Indeterminate dendritic cell
     * Primary MHN
     * Secondary to:
     * ALL
     * Follicular lymphoma
     * Other B-cell lymphoma
     * Other hematologic malignancy
     * Histiocytosis
  6. ALK-positive Histiocytosis
  7. Mixed Histiocytosis (MXH)
     * ECD/LCH
     * RDD/LCH
     * RDD/ECD
     * LCH/JXG
     * Other
  8. Other
     * Multicentric reticulohistiocytoma (MRH)
     * Necrobiotic xanthogranuloma (NX)
     * Not otherwise specified (NOS)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Collecting data on disease presentation, treatments used and treatment outcomes over time for patients diagnosed with RHD to better understand the diseases and optimize the treatments. | Data will be analysed on average yearly, the registry will be ongoing for 10 years.
  Collecting data on disease presentation, treatments used and treatment outcomes over time for patients diagnosed with RHD to better understand the diseases and optimize the treatments. Data will be analysed on average yearly, the registry will be ongoing for 10 years.

SECONDARY OUTCOMES:
Develop treatment guidelines for the RHD based on solid clinical trial data. | Data will be analysed on average yearly, the registry will be ongoing for 10 years.
  Develop treatment guidelines for the RHD based on solid clinical trial data. Data will be analysed on average yearly, the registry will be ongoing for 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Abla, MD, Principal Investigator — The Hospital for Sick Children
Locations (15):
- United States (6):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Hospital Nacional de Pediatria Garrahan, Buenos Aires, Argentina
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
- University Hospital Brno, Brno, Czechia
- Rostock University Medical Hospital, Rostock, Germany
- Azienda Ospedaliero-Universitaria Meyer, Florence, Italy
- Prinses Maxima Center, Utrecht, CS, Netherlands
- Children's Memorial Health Institute, Warsaw, Poland
- Hospital Universitario Cruces, Barakaldo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weitzman S, Jaffe R. Uncommon histiocytic disorders: the non-Langerhans cell histiocytoses. Pediatr Blood Cancer. 2005 Sep;45(3):256-64. doi: 10.1002/pbc.20246. PMID 15547923